CLINICAL TRIAL: NCT02608112
Title: Subcutaneous Tocilizumab in Monotherapy or in Combination With csDMARD in Patients With Moderate to Severe Active Rheumatoid Arthritis and Followed by Hospital and Office Based Rheumatologists: Non Interventional Study to Describe Real-World Drug Retention Rate of the Biotherapy at 1 Year
Brief Title: Study to Describe Real World Drug Retention Rate of the Tocilizumab at One Year
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29256
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with Moderate to Severe RA: Participants with moderate or severe RA, naïve to TCZ treatment (IV or SC), and who have no contra-indication to TCZ SC therapy as per the local label are included.
  Interventions: Drug: Methotrexate; Drug: Tocilizumab

INTERVENTIONS:
Drug: Methotrexate — Administered as per investigator's discretion. Investigator could also suggest any other csDMARDs instead of methotrexate.
Drug: Tocilizumab — Tocilizumab treatment will be administered SC at the discretion of the investigator in accordance with local clinical practice and local labelling.

SUMMARY:
This multicenter, prospective, non-interventional study is designed to obtain an accurate estimation of the drug retention rate of Tocilizumab (TCZ) Subcutaneously (SC) under real-world conditions in participants with moderate to severe rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Participants at least 18 years old
* Participants with moderate to severe RA not previously treated with TCZ (Intravenous [IV] or SC) for whom the rheumatologists have decided to initiate TCZ SC treatment as monotherapy or in combination with another conventional synthetic disease modifying anti-rheumatic drugs (csDMARD)

Exclusion Criteria:

* Participants taking part in a clinical trial on RA at the time of inclusion
* Participants with a contra-indication to TCZ SC therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe RA not previously treated with TCZ (IV or SC) for whom the rheumatologists have decided to initiate TCZ SC treatment as monotherapy or in combination with another csDMARD.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Estimated)
Dates: Start 2015-12-31 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Were on TCZ SC for a Period of 12 Months | Up to 12 Months

SECONDARY OUTCOMES:
Disease Activity Score Based on 28 Joints Count and C-Reactive Protein (DAS28-CRP) | Months 3, 6, 12, and 18
Simple Disease Activity Index (SDAI) | Months 3, 6, 12, and 18
Clinical Disease Activity Index (CDAI) | Months 3, 6, 12, and 18
Percentage of Participants With EUropean League Against Rheumatism (EULAR) Response | Months 3, 6, 12, and 18
Percentage of Participants Who Were on TCZ SC for a Period of 6 Months | Up to 6 Months
Percentage of Participants Who Were on TCZ SC for a Period of 18 Months | Up to 18 Months
Percentage of Participants who were on TCZ SC at 6, 12 and 18 Months Among 2 Subgroups: Participants Administered TCZ SC as Monotherapy and Participants Administered TCZ SC with Methotrexate or csDMARD | Up to 18 Months
Dose of Concomitant Steroids After Introduction of TCZ SC | Months 6, 12, and 18
Number of Participants with Adherence to TCZ SC Using the Compliance Questionnaire of Rheumatology 5 (CQR5) and Participants Diary Data | Months 6, 12, and 18
Percentage of Participants with Definitive Discontinuation of Treatment | Up to 18 Months
Percentage of Participants Performing All Visits at Hospital/Office Based Rheumatologist | Up to 18 Months
Percentage of Participants Taking Sick Leaves or Getting Hospitalized Due to RA | Up to 18 Months
Tender Joints Count | Months 3, 6, 12, and 18
Swollen Joints Count | Months 3, 6, 12, and 18
Disease Activity Score Based of 28 Joints Count and Erythrocyte Sedimentation Rate (DAS28-ESR) | Months 3, 6, 12, and 18

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (77):
- France (77):
  - Hopital Nord; Rhumatologie, Amiens
  - Ch D Ardeche Meridionale; Medecine A2, Aubenas
  - Ch De Belfort; Rhumatologie, Belfort
  - Institut Calot Helio Marin; Rhumatologie, Berck
  - Hopital Jean Minjoz, Besançon
  - Hopital Pellegrin; Rhumatologie, Bordeaux
  - Hopital La Cavale Blanche; Rhumatologie, Brest
  - Hopital Cote De Nacre; Rhumatologie, Caen
  - CH Jean Rougier; Rhumato Reed Fonctionnelle, Cahors
  - Infirmerie Protestante; Medecine interne Cancerologie, Caluire-et-Cuire
  - Hopital Pierre Nouveau;Medecine C Unite Rhumatologie, Cannes
  - Cabinet medical,Rhumatologie, Castelnaudary
  - Hopital Trousseau; Rhumatologie, Chambray-lès-Tours
  - HIA PERCY; Medecine Interne, Clamart
  - Hopital Gabriel Montpied; Service de Rhumatologie, Clermont-Ferrand
  - CH compiègne, Compiègne
  - Centre Hospitalier Alpes, Contamine-sur-Arve
  - Chu Sud Francilien; Rhumatologie, Corbeil-essones
  - CH Sud Francilien; Rhumatologie, Corbeil-Essonnes
  - Hopital Henri Mondor; Rhumatologie, Créteil
  - CH de Dax, Dax
  - Ch De Douai; Medecine Polyvalente, Dechy
  - Ch Louis Pasteur; Rhumato Med Interne Neurologie, Dole
  - Hopital Victor Jousselin; Rhumatologie 4EME Sud, Druex
  - Hopital Sud; Rhumatologie, Échirolles
  - Chi Alpes Du Sud Site De Gap; Med Interne Et Polyvalente, Gap
  - Cabinet Medical., Haguenau
  - Cabinet Medical, Haguenau
  - Cabinet medical; Rhumatologie, Joué-lès-Tours
  - CH de Juvisy sur Orge; Consult. externes, Juvisy-sur-Orge
  - Cabinet, La Madeleine
  - Hopital La Source; Rhumatologie, La Source
  - Ch De Laon; Medecine Interne, Laon
  - Ch Louis Pasteur; Medecine B3, Le Coudray
  - CH de Bicêtre; Rhumatologie, Le Kremlin-Bicêtre
  - Hopital Emile Roux; Rhumatologie, Le Puy-en-Velay
  - Hopital B Roger Salengro; Rhumatologie, Lille
  - Cabinet medical., Lille
  - Hopital Dupuytren; Rhumatologie, Limoges
  - Cabinet de Rhumatologie MSP de Beaublanc, Limoges
  - Ctre De Rhumato Lyon Presqu ile, Lyon
  - Hopital Edouard Herriot; Pavillon F Rhumatologie, Lyon
  - Hopital Sainte Marguerite; Rhumatologie, Marseille
  - Fondation Hopital Saint Joseph; Rhumatologie, Marseille
  - CH Annecy Genevois; Rhumatologie, Metz-Tessy
  - GHI Le Raincy Montfermeil, Montfermeil
  - Cabinet medical; Cabinet medical, Montpellier
  - Cabinet Medical, Montpellier
  - Hopital Lapeyronie; Immunologie Rhumatologie, Montpellier
  - Hôpital Lapeyronie; Immuno-Rhumatologie Pr Jorgensen, Montpellier
  - Ch Des Pays De Morlaix; Medecine I, Morlaix
  - Cabinet Medical, Nice
  - Hopital Pasteur; Rhumatologie, Nice
  - Maison de Santé; MSP, Nogent-le-Rotrou
  - Ch Pitie Salpetriere; Rhumatologie, Paris
  - Hopital De La Croix Saint Simon; Medecine Interne Rhumatologie, Paris
  - Ch Lyon Sud; Rhumato Secteur Jules Courmont, Pierre-Bénite
  - Cabinet, Poitiers
  - Chu La Miletrie; Rhumatologie, Poitiers
  - Hopital Sud Anne de Bretagne; Rhumatologie, Rennes
  - Hôpital Victor Provo, Roubaix
  - Centre Medico-Chirurgical de Touraine, Saint-Cyr-sur-Loire
  - Cabinet Medical, Saint-Lô
  - Hopital Instruction Armees Begin; Rhumatologie, Saint-Mandé
  - Centre Hopsitalier Saint Nazaire; Medecine Polyvalente, Saint-Nazaire
  - Hopital Nord; Rhumatologie, Saint-Priest-en-Jarez
  - Centre Hospitalier Saint Quentin, Saint-Quentin
  - CH de Saint Quentin, Saint-Quentin
  - Centre medical des coteaux; Rhumatologie, Saintes
  - Hopital Hautepierre; Rhumatologie, Strasbourg
  - Hopitaux du Leman site Thonon; Rhumatologie, Thonon-les-Bains
  - Cabinet de Rhumatologie, Toulouse
  - Hopital Purpan; Rhumatologie, Toulouse
  - Cabinet Medical, Tours
  - Cabinet Medical, Valenciennes
  - Hopitaux De Brabois; Rhumatologie, Vandœuvre-lès-Nancy
  - Hopital; Pole geriatrique, Villeneuve-sur-Lot

REFERENCES:
- [Derived] Hilliquin P, Barnetche T, Baillet A, Flipo RM, Lespessailles E, Roux C, Fardellone P, Gilbert-Marceau A, Idier I, Constantin A, Shipley E, Baudens G, Saraux A. Real-World 1-Year Retention Rate of Subcutaneous Tocilizumab Treatment in Patients with Moderate to Severe Active Rheumatoid Arthritis: TANDEM Study. Rheumatol Ther. 2021 Mar;8(1):95-108. doi: 10.1007/s40744-020-00253-0. Epub 2020 Nov 20. PMID 33216287